CLINICAL TRIAL: NCT05842993
Title: Efficacy and Safety of Hydrogen Inhalation in Subjects With Type 2 Diabetes
Brief Title: Study of Hydrogen Inhalation Compared With Placebo in Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Collaborators: Qingdao Hiser Medical Group (Other)
Responsible Party: Principal Investigator, Tongshang Ni, Lecturer, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QDU-HD-2023/1732
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes mellitus; hydrogen inhalation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen inhalation (Experimental): Patients receive hydrogen inhalation.
  Interventions: Device: Hydrogen generator
- Placebo (Placebo Comparator): Patients receive placebo.
  Interventions: Device: Analogue machine

INTERVENTIONS:
Device: Hydrogen generator — Patient inhales hydrogen gas for 2 hours per day in the flow rate of 2L/min via nasal cannula by applying hydrogen generator (HZS-2700A, Qingdao Haizhisheng Corp.,LTD, Qingdao, China) for 12 weeks.
  Arms: Hydrogen inhalation
Device: Analogue machine — Patient inhales normal air for 2 hours per day in the flow rate of 2L/min via nasal cannula with analogue machine for 12 weeks. This machine has the same appearance as the hydrogen generator.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hydrogen inhalation in type 2 diabetes patients.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy and safety of hydrogen inhalation compared with placebo in patients with type 2 diabetes mellitus after 12-week treatment in a randomized, double-blind, placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old and gender of both sex;
2. Body mass index 18.5kg/m2 to 40 kg/m2;
3. Diagnosed as type 2 diabetes according to the diagnostic criteria of type 2 diabetes established by WHO in 1999;
4. Patients with type 2 diabetes whose blood glucose is not well controlled after diet control and exercise therapy for more than 3 months;
5. HbA1c 7% to 10%, and fasting venous plasma glucose ≤ 15 mmol/L;
6. Be able to understand the procedures and methods of this clinical study, voluntarily participate in and sign the informed consent.

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, or other specific types of diabetes;
2. Screening for having received anti-diabetic drug therapy within 3 months or receiving continuous anti-diabetic drug therapy at any time before screening for more than 3 months;
3. History of diabetic ketoacidosis, diabetic hyperglycemic hyperosmolar syndrome, lactic acidosis, diabetic hypoglycemia; or is currently combined with retinopathy, diabetic nephropathy and diabetic neuropathy;
4. Hyperlipidemia patients with irregular or unstable dose of lipid-lowering drugs
5. Chronic gastrointestinal disorders with obvious digestive and absorption disorders, as well as other endocrine diseases, such as hyperthyroidism, hypercortisolism, acromegaly, etc.;
6. Patients with diseases that may worsen due to intestinal flatulence (such as Roemheld syndrome, severe hernia, intestinal obstruction, intestinal surgery and intestinal ulcers);
7. Had transient ischemic attack, cerebrovascular accident or unstable angina in the past 6 months; History of myocardial infarction or had conducted coronary angioplasty or coronary artery bypass graft surgery; Heart failure (NYHA classification Stage III or IV), or left ventricular hypertrophy indicated by ECG;
8. Subjects (taking or not taking antihypertensive drugs) had poor blood pressure control (SBP ≥ 160mmhg, or DBP ≥ 100mmhg);
9. liver disease, ALT or AST > 2 ULN, or TBIL > 2 ULN, and the diagnosis was confirmed within one week;
10. Patients with renal function impairment (Cr > 1 ULN or Ccr < 60ml / min) and confirmed by reexamination within one week;
11. Had malignancy in the past 5 years, not including basal cell carcinoma;
12. History of acute or chronic pancreatitis, or related diseases that are most common cause of acute pancreatitis (such as recurrent cholelithiasis, etc.);
13. Combined use of drugs that affect glucose metabolism, such as glucocorticoids;
14. Combined use of Chinese herbal medicine with the effect of regulating blood glucose within 3 months;
15. Those who have serious diseases and may be in danger of life during treatment and follow-up;
16. Mental and neurological disorders, unable to correctly express their wishes;
17. Alcoholics and drug abusers and addicts;
18. Women of childbearing age are pregnant, breastfeeding, have pregnancy intentions or have a positive pregnancy test (urine HCG or blood HCG), and should not take effective contraceptive measures during the trial (effective contraceptive measures include sterilization, intrauterine device, oral contraceptive or diaphragm method prescribed by local law);
19. Patients who have participated in clinical trials of other drugs or medical devices in the past 3 months;
20. Patients with other diseases that the researchers believe will not be able to evaluate or are unlikely to complete the expected course of treatment and follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) | Baseline and Week 12
  The change in HbA1c from baseline to Week 12 in hydrogen inhalation group compared to Placebo.

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG) | Baseline and Week 12
  The change in FPG from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in 2h-postprandial plasma glucose (2h-PPG) | Baseline and Week 12
  The change in 2h-PPG from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Patients with HbA1c <7.0% | At Week 12
  Percentage of patients reaching HbA1c <7% at Week 12
Patients with HbA1c <6.5% | At Week 12
  Percentage of patients reaching HbA1c <6.5% at Week 12
Change in fasting plasma insulin | Baseline and Week 12
  The change in fasting plasma insulin from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in insulin sensitivity and beta cell function assessed by the homeostatic model assessment (HOMA) | Baseline and Week 12
  The change in HOMA-IR and HOMA-β from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in serum lipid profile | Baseline and Week 12
  The change in total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in waist circumference | Baseline and Week 12
  The change in waist circumference from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in body weight | Baseline and Week 12
  The change in body weight from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in body mass index (BMI) | Baseline and Week 12
  The change in BMI from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in blood pressure | Baseline and Week 12
  The change in blood pressure from baseline to Week 12 in hydrogen inhalation group compared to Placebo.
Change in oxidative stress index and inflammatory index | Baseline and Week 12
  Serum MDA and SOD, TNF-α, IL-6 quantifications were conducted using commercial kits from baseline to Week 12.
Safety measurement | Baseline to Week 12
  The incidence rates of adverse events, clinical findings in the physical examination, vital signs, 12-lead electrocardiogram (ECG), clinical laboratory tests (hematology, blood biochemistry, and urinalysis) from baseline to Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Tongshang Ni, Ph.D, Principal Investigator — Qingdao University
Locations (1):
- Qingdao Traditional Chinese Medicine Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No